CLINICAL TRIAL: NCT02807389
Title: A Phase I Study of Autologous Mesenchymal Stromal Cell Coated Fistula Plug in Patients With Complicated Post-surgical Fistulas
Brief Title: Stem Cell Fistula Plug in Post Surgical Leak Fistulas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William A. Faubion, M.D., MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-004326
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Surgical Leak Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MSC Fistula plug: Single Treatment Group (Experimental): All patients received treatment of a stem cell coated fistula plug.
  Interventions: Drug: MSC Fistula Plug

INTERVENTIONS:
Drug: MSC Fistula Plug — Eligible patients will be treated with a fistula plug that has been coated with autologous mesenchymal stromal cell.
  Other Names: mesenchymal stromal cell coated fistula plug

SUMMARY:
The investigators propose to study the safety of autologous mesenchymal stromal cell transfer using a biomatrix (The Gore Fistula Plug) in a Phase I study using a single dose of 20 million cells. 15 adult patients (age 18 and greater) with persistent symptomatic post-surgical gastrointestinal leaks despite current standard radiologic and endoscopic therapies will be enrolled. The subjects will be subsequently followed for fistula response and closure for 18 months. This is an autologous product derived from the patient and used only for the same patient.

DETAILED DESCRIPTION:
Visit 1: Patients will be evaluated for eligibility (inclusion/exclusion checklist) and written, informed consent will be obtained. Patients will undergo general exam with vital signs. Patients will be scheduled for a fat biopsy to collect the tissue needed to grow MSC. In the event there is no cell growth from the tissue obtained from the first biopsy, one further attempt will made from a second tissue sample from this patient. However, if the second attempt fails to grow cells, no further attempts will be made, and the subject will not continue in the study.

Visit 2 (Week 0; Day 0): Patients will undergo an interventional endoscopy, the fistula tract will be assessed and the stem cell coated will be placed endoscopically.

Study visit will be as follows:

Visit 3 (Week 0; Day 1) Visit 4 (Week 2; Month 1) Visit 5 (Week 4; Month 1) Visit 6 (Week 8; Month 2) Visit 7 (Week 12; Month 3) Visit 8 (Week 24; Month 6) Visit 9 (week 52; Month 12) Visit 10 (Week 78; Month 18)

ELIGIBILITY:
Inclusion Criteria

1. Males and females 18-75 years of age.
2. Residents of the United States.
3. Patients with persistent symptomatic fistulas arising after gastro-esophageal resections, enteric or colonic resections or Bariatric surgeries.
4. Single-tract fistula
5. Have no contraindications to imaging evaluations: e.g. contrast allergies
6. Ability to comply with protocol
7. Competent and able to provide written informed consent
8. Must have failed standard conservative therapy which includes at least one endoscopic attempt to resolve fistula. Standard conservative management includes drainage of sepsis, antibiotics, nutritional support, etc. Endoscopic closure attempt with devices such as, but not limited to; endo-stitch, clipping, surgical sealants, etc. This attempt may be with or without diversion of the luminal contents by stenting.
9. Radiographic Imaging within 7 days of fistula plug placement (e.g. CT, PET, etc.).

Exclusion Criteria

1. Inability to give informed consent.
2. Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
3. Specific exclusions;

   a. Evidence of hepatitis B, C, or HIV
4. Investigational drug within thirty (30) days of baseline
5. A resident outside the United States
6. History of clinically significant auto-immunity (i.e. Inflammatory Bowel Disease).
7. Previous allergic reaction to a fistula plug.
8. If obtaining sufficient adipose tissue for manufacturing is not technically feasible
9. Allergic to local anesthetics
10. Pregnant patients or trying to become pregnant or breast feeding.
11. Non-enterocutaneous tracts
12. Fistula output >2000 ml/day
13. Multiple or end fistulas
14. Fistulous tract <2 cm in length
15. Fistulous tract or defect >1 cm in diameter,
16. Fistulas opening into abdominal wall defect.
17. Diseased adjacent bowel, fistula in the radiation field, persistent distal obstruction or malignancy
18. Patients on immunosuppression or chemotherapy
19. Uncontrolled diabetes, i.e. blood sugar more than 200
20. Sepsis
21. Fistulas arising from a malignant lesion
22. Patients with obstructive malignancies
23. Patients with stage III and/or stage IV cancers. The investigators will exclude patients with stage III or IV cancers, poorly differentiated cancers and patients with less than accepted disease free surgical margins.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2-18 months
  Data collection will include: worsening of the fistula, abnormal laboratory values, or significant abnormalities in physical examination. The Outcome Measure will be the number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

SECONDARY OUTCOMES:
Incidence of Fistula Closure | 2-18 months
  Data collection will include: degree of drainage cessation from fistula. The Outcome Measure will be the number of Participants With Closure of their Fistula.

CONTACTS AND LOCATIONS:
Overall Officials: William A Faubion, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials